CLINICAL TRIAL: NCT04872231
Title: A Randomized, Double-Blind, Placebo Controlled, Single-Dose and Multiple Dose Dose-Ranging Study of Voriconazole Inhalation Powder in Healthy Adult Subjects
Brief Title: Single Ascending Dose and Multiple Ascending Dose Study of Voriconazole Inhalation Powder in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TFF Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: TFF-V1-001
Record Dates: First submitted 2021-04-29; First posted 2021-05-04 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Healthy
Keywords: voriconazole; inhaled; VFEND; aspergillosis; IPA; fungal infection; pulmonary aspergillosis
MeSH Terms: conditions — Respiratory Aspiration; Aspergillosis; Mycoses; Pulmonary Aspergillosis

STUDY DESIGN:
Intervention Model Description: Part A: Eight (8) subjects will participate in each of the 4 dose escalations. Subjects will be randomized to receive either Voriconazole Inhalation Powder or placebo by inhalation (6 active, 2 placebo per group of 8).
  Part B: Eight (8) subjects will participate in each of the 4 dose escalations. Subjects will be randomized to receive either Voriconazole Inhalation Powder or placebo by inhalation (6 active, 2 placebo per group of 8).
Who Masked: Participant, Investigator
Masking Description: The investigators, study coordinators, study subjects and the Sponsor will be blinded to treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Voriconazole Inhalation Powder (Experimental): Investigational drug will be supplied as capsules, each capsule contains 10 mg of Voriconazole Inhalation Powder. The capsules will be administered with the provided breath actuated Plastiape RS00 Model 8 Dry Powder Inhaler device.
  Interventions: Drug: Voriconazole Inhalation Powder
- Placebo (Placebo Comparator): Placebo will be supplied as capsules, each capsule will contain no active ingredient. The capsules will be administered with the provided breath actuated Plastiape RS00 Model 8 Dry Powder Inhaler device.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Voriconazole Inhalation Powder — PART A (SAD): Voriconazole Inhalation Powder (VIP) will be supplied as one to eight 10 mg capsules. Each capsule contains 10 mg of VIP and will be administered with a Plastiape RS00 Dry Powder inhaler. Doses may require multiple inhalations. All inhalations must be conducted within a 10-minute period.
  SAD subjects will receive a single dose of study medication. Subjects in Cohort 1 will receive 10 mg, Cohort 2: 20 mg, Cohort 3: 40 mg, Cohort 4: 80 mg.
  PART B (MAD): Voriconazole Inhalation Powder (VIP) and will be administered with a will be supplied as one to eight 10 mg capsules. Each capsule contains 10 mg of VIP and will be administered with a Plastiape RS00 Dry Powder inhaler. Doses may require multiple inhalations. All inhalations must be conducted within a 10-minute period.
  MAD subjects will receive VIP BID for a total of 13 doses. Subjects in Cohort 1 will receive 10 mg BID, Cohort 2: 20 mg BID, Cohort 3: 40 mg BID, Cohort 4: 80 mg BID.
  Other Names: VIP
  Arms: Voriconazole Inhalation Powder
Drug: Placebo — PART A (SAD): Placebo capsules will be supplied as one to eight capsules. Each capsule contains placebo inhalation powder. The capsules will be matched for use within the provided Plastiape RS00 Dry Powder inhaler device (Model 8). Doses may require multiple inhalations through the inhaler device. All inhalations must be conducted within a maximum of 10-minute period.
  Subjects in PART A will receive a single dose of placebo.
  PART B (MAD): Placebo will be supplied as one to eight capsules. Each capsule contains placebo inhalation powder. The capsules will be matched for use within the provided Plastiape RS00 Dry Powder inhaler device (Model 8). Doses may require multiple inhalations through the inhaler device. All inhalations must be conducted within a maximum of 10-minute period.
  Subjects in PART B will receive Placebo BID for a total of 13 doses.
  Other Names: Vehicle
  Arms: Placebo

SUMMARY:
This is a Phase 1 (healthy adult volunteers), 2-part, double-blind, randomized, placebo controlled trial to evaluate the safety and pharmacokinetic (PK) profiles of escalating single doses of Voriconazole Inhalation Powder versus placebo (SAD part) and escalating multiple doses of Voriconazole Inhalation Powder versus placebo (MAD part). SAD part will be initiated first and includes a sentinel design. MAD part will not utilize a sentinel design and will be initiated once the lowest doses from SAD part are deemed safe.

DETAILED DESCRIPTION:
This is a Phase 1, randomized, 2 part double-blind, placebo-controlled trial to evaluate the safety and PK profiles of Voriconazole Inhalation Powder (VIP) in a SAD/MAD study design.

Part A is a double-blinded, placebo-controlled, randomized, dose- ranging single dose study evaluating four different dose levels.

On Day 1 of each group, two selected subjects (sentinel subjects) will receive either Voriconazole Inhalation Powder or a matching placebo. Blood and sputum samples and safety measurements including Adverse Events (AEs) will be collected over 24 hour period following the drug administration. The safety results to be evaluated include AEs, concomitant medications, out of specification clinical laboratory results, vital signs, Electrocardiograms (ECGs), visual examinations, pulmonary function tests, pulse oximetry results and any new findings on physical examinations. If the administration is safe as deemed by Principal Investigator & Medical Monitor, the remaining six subjects will be dosed, with identical safety and PK procedures performed after minimum of 3 days interval. A minimum of 3 days will separate each dose escalation, with the remaining dose groups dosed in a sentinel fashion.

Part B is a double-blinded, placebo-controlled, randomized, dose- ranging multi-dose study evaluating four different dose levels. Dose level 1 of Part B can begin in parallel once safety assessments of Part A dose level 2 are complete and indicate safety is present. Voriconazole Inhalation Powder will be administered twice daily (BID) × 13 doses. Blood samples for safety and PK will be collected over 12 hours after the first dose and 24 hours after the last dose. A minimum of 1 week will separate the start of each dose escalation, with the remaining dose groups.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent to participate.
2. Healthy, adult males or females (women of non-childbearing potential only).
3. Body mass index (BMI) ≥ 18.0 and ≤ 32.0 kg/m2 at Screening.
4. Medically healthy with no clinically significant abnormalities in medical history, physical and visual examination, laboratory profiles, vital signs or ECGs, as deemed by the PI or designee.
5. Agree to abstain from recreational drug use throughout the study.
6. Must be willing and able to comply with the protocol.
7. Succeed in training on the use of the device for maximum of 12 inhalations in total, with demonstration of at-least 8 successful inhalations of empty capsules during training.
8. Have had a forced expiratory volume in one second (FEV1) ≥80%.

Exclusion Criteria:

1. Is mentally or legally incapacitated or has significant emotional problems in the opinion of the PI.
2. History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the PI.
3. History of any illness that, in the opinion of the PI, might confound the results of the study or poses an additional risk to the subject by their participation in the study.
4. History or presence of alcoholism or drug abuse within the past 2 years.
5. History or presence of hypersensitivity or idiosyncratic reaction to voriconazole or any triazole antifungal.
6. Has had surgery or any medical condition within 6 months prior to first dosing which may affect the absorption, distribution, metabolism, or elimination of the study drug, in the opinion of the PI or designee.
7. Female subjects of childbearing potential.
8. Female subjects with a positive pregnancy test or who are lactating.
9. Positive urine drug or alcohol results at screening or first check-in.
10. Positive cotinine results at screening.
11. Diagnosis of asthma.
12. Use of albuterol or a similar bronchodilator
13. Positive results at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV).
14. QTcF interval is >450 msec or has ECG findings deemed abnormal with clinical significance by the PI at screening.
15. Seated blood pressure with systolic less than 90 mmHg or diastolic less than 60 mm/Hg or with a systolic greater than 140 mmHg or diastolic greater than 90 mmHg at screening.
16. Seated heart rate is lower than 60 bpm or higher than 100 bpm at screening.
17. Using any exclusionary medication.
18. Donation or loss of 50 to 499 mL whole blood within 30 days or more than 499 mL whole blood within 56 days prior to the first dosing.
19. Plasma donation within 7 days prior to the first dosing.
20. Has coagulation test outside of normal ranges.
21. Has platelet, hemoglobin, and hematocrit that are below the lower limit of normal.
22. Has liver function tests including alanine aminotransferase (ALT), aspartate aminotransferase (AST), ALP and total bilirubin that are greater than the upper limit of normal. Estimated creatinine clearance <90 mL/min at screening.
23. Participation in another clinical study within 30 days prior to the first dosing.
24. Had a treatment with other investigational drug within 5 times the elimination half- life, if known (e.g., a marketed product) or within 30 days (if the elimination half-life is unknown) prior to first dosing.
25. Demonstrates an inability to operate the inhalation device after training.
26. Allergy or sensitivity to lactose or milk products.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2019-11-22 (Actual); Primary Completion 2020-07-29 (Actual); Study Completion 2020-08-26 (Actual)

PRIMARY OUTCOMES:
Number of participants who experience Adverse Events (AEs), Serious Adverse Events (SAEs) and withdrawals due to AEs | Through study completion, an average of 14 days
  Number of AEs, SAEs, and discontinuations due to AEs
Number of participants who experience vital sign abnormalities | Baseline through study completion, an average of 14 days
  Number of participants with potentially clinically significant vital sign values
Number of participants who experience pulse oximetry abnormalities | Baseline through study completion, an average of 14 days
  Number of participants with potentially clinically significant pulse oximetry values
Mean change from baseline in forced expiratory volume (FEV1) | Baseline through study completion, an average of 14 days
  Spirometry used to measure FEV1 lung function
Mean change from baseline in forced vital capacity (FVC) | Baseline through study completion, an average of 14 days
  Spirometry used to measure FVC lung function
Mean change from baseline in FEV1/FVC ratio | Baseline through study completion, an average of 14 days
  Spirometry used to measure FEV1 and FVC lung function
Mean change from baseline in QTcF changes via ECG | Baseline through study completion, an average of 14 days
  Number of participants with potentially clinically significant ECG values
Number of participants who experience physical examination abnormalities | Baseline through study completion, an average of 14 days
  Number of participants with potentially clinically significant physical examination findings
Number of participants who experience laboratory test abnormalities | Baseline through study completion, an average of 14 days
  Number of participants with potentially clinically significant laboratory test results
PK of VIP in plasma: Area under the plasma-concentration time curve (AUC) | Predose Day 1 and through 12 hours post last dose (day 6)
  Blood samples will be collected for plasma analysis
PK of VIP in plasma: Area under the concentration time curve, from time 0 to the last observed non-zero concentration (AUC0-tlast) | Predose Day 1 and through 12 hours post last dose (day 6)
  Blood samples will be collected for analysis
PK of VIP in plasma: Maximum observed concentration (Cmax) | Predose Day 1 and through 12 hours post last dose (day 6)
  Blood samples will be collected for analysis
PK of VIP in plasma: Time to maximal observed concentration (tmax) | Predose Day 1 and through 12 hours post last dose (day 6)
  Blood samples will be collected for analysis
PK of VIP in plasma: Area under the plasma-concentration time curve over the first 12 hours after dosing (AUC0-12) | Predose Day 1 and through 12 hours post last dose (day 6)
  Blood samples will be collected for analysis
PK of VIP in plasma: Area under the concentration time curve from time 0 extrapolated to infinity (AUC∞) | Predose Day 1 and through 12 hours post last dose (day 6)
  Blood samples will be collected for analysis
PK of VIP in plasma: Termination elimination half-life (t½) | Predose Day 1 and through 12 hours post last dose (day 6)
  Blood samples will be collected for analysis
PK of VIP in plasma: Apparent total body clearance (CL/F) | Predose Day 1 and through 12 hours post last dose (day 6)
  Blood samples will be collected for analysis
PK of VIP in plasma: Apparent volume of distribution during the terminal elimination phase (Vz/F) | Predose Day 1 and through 12 hours post last dose (day 6)
  Blood samples will be collected for analysis

CONTACTS AND LOCATIONS:
Overall Officials: Dale Christensen, PhD, Study Director — TFF Pharmaceuticals
Locations (1):
- Cliantha Research, Mississauga, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No